CLINICAL TRIAL: NCT00890292
Title: An Open-Label, Multi-Center, Sequential Group, Ascending Dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of JNJ-31001074 After a Single Dose Administration in Pediatric Subjects With Attention-Deficit/Hyperactivity Disorder, 12 to 17 Years Old
Brief Title: A Study to Evaluate Pharmacokinetics, Safety and Tolerability After a Single Dose Administration of JNJ-31001074 in Pediatric Patients (12-17 Years) With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Clinical Leader Psychiatry, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR016186
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Attention Deficit Hyperactivity Disorder; Attention Deficit Disorders With Hyperactivity
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; JNJ-31001074
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — bavisant

INTERVENTIONS:
Drug: JNJ-31001074

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (process by which JNJ-31001074 is absorbed, distributed, metabolized, and eliminated by the body) after a single dose of JNJ-31001074. Up to three dose strengths will be tested in patients 12-17 years old with attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
This will be an open-label (both the physician and patient know which treatment will be administered), multicenter, sequential-group (one group after another), single-dose, Phase I study in 12-17 year old patients with attention deficit hyperactivity disorder (ADHD). Patients in the first group will be administered a single dose of JNJ-31001074 while they are observed and tested (blood and urine samples collected) for a period of time. If they do not exhibit any adverse side effects and the data collected is within the predicted safe values, the dose will be increased for a new group of patients. Three dose groups are planned (0.015, 0.045 and 0.15 mg/kg) and up to 18 patients will complete the study.The study consists of a screening phase, an open-label treatment phase, and an end-of-study/early withdrawal assessments. During screening, patients will be required to give their assent to participate (agreement to participate) in the study and parents/guardians will be required to provide their consent. Patients will be evaluated to see if they meet selection criteria specified in the protocol. Patients who meet the selection criteria at screening will report to the study center on the evening prior to Day 1 to confirm that they continue to meet the eligibility requirements. If the patient is still eligible, they will be admitted to the study center and will be required to fast (no food or beverages) for at least 4 hours prior to their dose. On Day 1, a single dose of either 0.015, 0.045 or 0.15 mg/kg of JNJ-31001074 will be administered at approximately 8 am, followed by multiple blood sampling and urine collection. At the Investigator's discretion, patients may be discharged on Day 3 after the last blood and urine samples are taken, or alternatively, they may be discharged on Day 1 after the 12-hour blood and urine samples are taken. In the latter case, patients will be required to return to the study center on Day 2 and Day 3 for additional blood and urine samples. Parent(s) may remain at the study center with their child. Patients in the first dose group of the study will receive a single 0.015 mg/kg dose of JNJ-31001074. The data obtained from the patients in the first dose group will be reviewed prior to the second dose group (0.045 mg/kg) being started. Data obtained from the patients in the second dose group will be reviewed prior to the third dose group (0.15 mg/kg) being started. All patients will be required to return to the study site for an end of study / early withdrawal assessment. The maximum duration of participation for each patient is expected to be 24 days. Depending on their body weight and which dose group they are participating in (0.015 mg/kg, 0.045 mg/kg or 0.15 mg/kg), patients will be dosed once with a combination of 0.25, 1, 3, and 5 mg tablets of JNJ-31001074 administered orally.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls with a Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) diagnosis of ADHD
* Height and weight within the 5th to 95th Physical Growth National Center for Health Statistics percentiles for age and sex
* Clinically stable with no changes in the management of ADHD for at least 1 week prior to screening
* Clinical Global Impression of Severity of Illness (CGI-S) score must be 3 or less at screening
* Children who are capable of providing assent (typically 7 years of age and older) must sign an assent form

Exclusion Criteria:

* History of or current clinically significant medical illness
* DSM-IV diagnosis of psychiatric disorder other than ADHD
* Have taken methylphenidate, amphetamine, or other stimulant medications within 5 half-lives before screening or atomoxetine within 30 days of screening
* Use of any prescription or nonprescription medication except for acetaminophen within 14 days before planned dosing of the study drug
* Positive test for drugs of abuse

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to evaluate the pharmacokinetics, safety, and tolerability of JNJ-31001074 after a single dose administration of JNJ-31001074 in pediatric patients with ADHD, 12 to 17 years of age, inclusive. | 3 days of blood and urine sampling

SECONDARY OUTCOMES:
Incidence and type of adverse events and changes in clinical laboratory results, electrocardiograms(ECGs),physical examination,vital signs,Clinical Global Impression of Severity of Illness(CGI-S) scale and Columbia-Suicide Severity Rating Scale (C-SSRS) | 24 days (includes a 21 day screening phase and a 3 day open-label treatment phase)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.